CLINICAL TRIAL: NCT04147403
Title: Xinhua Hospital, Affiliated to Shanghai Jiao Tong University, School of Medicine
Brief Title: A Study of Extended Total Mesopancreas Excision(eTME) for Pancreatic Head Adenocarcinoma.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Yingbin Liu, MD, PhD, FACS, Prof., Shanghai Jiao Tong University School of Medicine
Other Study IDs: ETMEFP_LYB_2019
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Pancreas Adenocarcinoma
Keywords: pancreatic head adenocarcinoma; total mesopancreas excision;pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study of extended total mesopancreas excision(eTME) for pancreatic head adenocarcinoma is a retrospective multicenter cohort, collecting medical records and follow-up data of patients who underwent radical resection with pancreatic head adenocarcinoma.

DETAILED DESCRIPTION:
The objectives of the study are as follows:

1. To evaluate the perioperative safety of extended total mesopancreas excision(eTME) for patients who diagnosed with resectable pancreatic head adenocarcinoma.
2. To demonstrate the prognosis of extended total mesopancreas excision(eTME) for patients who diagnosed with resectable pancreatic head adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pancreatic head adenocarcinoma who underwent curative-intent resection.
2. Patients with accessible medical records

Exclusion Criteria:

1. Patients with unknown chemotherapy sequence or status
2. Patients with history of previous malignant tumors
3. Patients with distant metastases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with resectable pancreatic head adenocarcinoma who underwent radical resection between January 1st 2008 and October 31st 2018 in collaborated tertiary hospital hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  The overall survival data were defined by (date of death)-(date of first diagnosis).The survival status of patients were retrieved from follow-up.

SECONDARY OUTCOMES:
Disease free survival | 5 years
  The overall survival data were defined by (date of recurrence/progression)-(date of surgery).During follow-up period, abdominal enhanced CT, chest X-ray, tumor markers and routine blood tests were carried out to evaluate recurrence/progression.

CONTACTS AND LOCATIONS:
Overall Officials: Yingbin Liu, Ph.D., Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (4):
- China (4):
  - Ruijin Hospital,Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Changhai Hospital Affiliated to Naval Medical University, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Affiliated to Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No